CLINICAL TRIAL: NCT01419171
Title: OMEGA: A Prospective, Multicenter Single-Arm Trial to Assess the OMEGA™ Coronary Stent System for the Treatment of a Single De Novo Coronary Artery Lesion
Brief Title: The OMEGA Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2215
Record Dates: First submitted 2011-08-16; First posted 2011-08-18 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Atherosclerosis; Coronary Artery Disease
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OMEGA™ Monorail Coronary Stent System (Experimental)
  Interventions: Device: OMEGA™ Monorail Coronary Stent System

INTERVENTIONS:
Device: OMEGA™ Monorail Coronary Stent System — All enrolled patients are treated with the OMEGA™ Monorail Bare Metal Coronary Stent System and followed for 12 months post-procedure.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the OMEGA Coronary Stent System for the treatment of subjects with a de novo atherosclerotic coronary artery lesion.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age.
* Subject (or legal guardian) indicates understanding of the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed.
* Subject is eligible for percutaneous coronary intervention (PCI).
* Subject has symptomatic coronary artery disease or documented silent ischemia.
* Subject is an acceptable candidate for coronary artery bypass grafting (CABG).
* Subject has a left ventricular ejection fraction (LVEF) ≥30% as measured within 60 days prior to enrollment.
* Subject is willing to comply with all protocol-required follow-up evaluations.

Angiographic Inclusion Criteria:

* Target lesion must be a de novo lesion located in a native coronary artery with a visually estimated reference vessel diameter (RVD) ≥ 2.25 mm and ≤4.5 mm.
* Target lesion length must measure (by visual estimate) as follows:

  * ≤28 mm for stent diameter lengths of 2.75 mm, 3.00 mm, 3.50 mm, 4.00 mm and 4.50 mm
  * ≤24 mm for stent diameter lengths of 2.25 mm and 2.50 mm
* Target lesion must be in a major coronary artery or branch with visually estimated stenosis ≥50% and <100% with Thrombolysis in Myocardial Infarction (TIMI) flow >1.
* Target lesion must be successfully pre-dilated.

Exclusion Criteria:

* Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute myocardial infarction (MI).
* Subject with unstable angina or recent MI (clinically diagnosed within 3 days) must have creatine kinase (CK)/ creatine kinase-myoglobin band(CK-MB) or troponin documented prior to the procedure and are excluded if any of the following criteria are met at the time of the index procedure:

  1. If CK MB >2× upper limit of normal (ULN), the subject is excluded regardless of the CK Total.
  2. If CK Total >2× ULN, CK-MB must be drawn and the subject is excluded if CK-MB is abnormal.
  3. If CK/CK-MB results are not available at the time of procedure, the subject is excluded if troponin >1× ULN and the subject has at least one of the following:

     * Subject has ischemic symptoms and ECG changes indicative of ongoing ischemia (e.g., >1 mm stent thrombosis (ST) segment elevation or depression in consecutive leads or new left bundle branch block [LBBB])
     * Development of pathological Q waves in the ECG or;
     * Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality Note: Subjects who do not have unstable angina or recent MI must still have CK/CK-MB drawn prior to the index procedure. However, the results for these subjects do not need to be available prior to the index procedure and there are no exclusion criteria based on these studies.
* Subject is receiving chronic (≥72 hours) anticoagulation therapy (e.g., heparin, coumadin) for indications other than acute coronary syndrome.
* Subject has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3.
* Subject has a white blood cell (WBC) count <3,000 cells/mm3.
* Subject has documented or suspected liver disease, including laboratory evidence of hepatitis.
* Subject is on dialysis or has known renal insufficiency (e.g. serum creatinine level >2.0 mg/dL).
* Subject has active peptic ulcer disease, an active gastrointestinal (GI) bleed, other bleeding diathesis or coagulopathy or will refuse transfusions.
* Subject has had a cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months, or has any permanent neurologic defect that may cause non-compliance with the protocol.
* Target vessel (including side branches) has been treated with any type of PCI (e.g., balloon angioplasty, stent, cutting balloon, atherectomy) within 12 months prior to the index procedure.
* Target vessel has been treated within 10 mm proximal or distal to the target lesion (by visual estimate) with any type of PCI (e.g., balloon angioplasty, stent, cutting balloon, or atherectomy) at any time prior to the index procedure.
* Non-target vessel or side branch has been treated with any type of PCI (e.g., balloon angioplasty, stent, cutting balloon, atherectomy) within 1 day prior to the index procedure.

Note: 1 lesion in a non-target vessel may be treated during the index procedure prior to the treatment of the target (study) lesion.

* Planned or actual target vessel treatment with an unapproved device, directional or rotational coronary atherectomy, laser, cutting balloon, or transluminal extraction catheter immediately prior to stent placement.
* Planned PCI or CABG after the index procedure.
* Subject previously treated at any time with coronary intravascular brachytherapy.
* Subject has known allergy to the study stent system or protocol-required concomitant medications (e.g., stainless steel, platinum, chromium, nickel, iron, thienopyridines and acetylsalicylic acid (ASA)) and contrast (that cannot be adequately premedicated).
* Subject has any other serious medical illness (e.g., cancer, congestive heart failure) that may reduce life expectancy to less than 12 months.
* Subject has current problems with substance abuse (e.g., alcohol, cocaine, heroin, etc.).
* Subject has a planned procedure that may cause non-compliance with the protocol or confound data interpretation.
* Subject is participating in another investigational drug or device clinical trial that has not reached its primary endpoint or intends to participate in another investigational drug or device clinical trial within 12 months after the index procedure.
* Subject is female of childbearing potential with a positive pregnancy test within 14 days before the index procedure, is lactating, or intends to become pregnant during the study.
* Subject has more than 1 target lesion, or more than 1 target lesion and 1 non-target lesion, which will be treated during the index procedure.

Angiographic Exclusion Criteria:

* Target lesion meets any of the following criteria:

  * Aorto-ostial location (i.e., lesion located within 5 mm of the ostium by visual estimate)
  * Left main location
  * Located within 5 mm of the origin of the left anterior descending (LAD) coronary artery or left circumflex (LCX) coronary artery or Right Coronary Artery (RCA) by visual estimate
  * Located within a saphenous vein graft or an arterial graft
  * Will be accessed via a saphenous vein graft or an arterial graft
  * Involves a side branch ≥2.0 mm in diameter by visual estimate
  * Involves a side branch <2.0 mm in diameter by visual estimate that has a clinically significant stenosis at the ostium
  * TIMI flow 0 (total occlusion) or TIMI flow 1 prior to guide wire crossing
  * Excessive tortuosity proximal to or within the lesion
  * Extreme angulation proximal to or within the lesion
  * Target lesion and/or target vessel proximal to the target lesion is moderately to severely calcified by visual estimate
  * Restenotic from previous intervention
  * Thrombus, or possible thrombus, present in the target vessel
  * Target lesion cannot be covered by a single study stent (unplanned bailout stenting is allowed)
* Non-target lesion to be treated during the index procedure meets any of the following criteria:

  * Located within the target vessel
  * Located within a bypass graft (venous or arterial)
  * Left main location
  * Chronic total occlusion
  * Involves a complex bifurcation (e.g., bifurcations requiring treatment with more than 1 stent)
  * Requires additional unplanned stents (treatment of the non-target lesion with more than one stent is permitted as long as the stents are initially planned)
  * Treatment not deemed a clinical angiographic success
  * Treatment not completed prior to treatment of target lesion
* Subject has unprotected left main coronary artery disease (>50% diameter stenosis).
* Subject has protected left main coronary artery disease and a target lesion in the LAD or LCX.
* Subject has an additional clinically significant lesion(s) in the target vessel for which an intervention within 12 months after the index procedure may be required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Maurer, MPH, Study Director — Boston Scientific Corporation
Locations (37):
- United States (22):
  - National Park Medical Center, Hot Springs, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Florida Hospital, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Southern Illinois University-Memorial Medical Center, Springfield, Illinois
  - St. Vincent's Hospital, Indianapolis, Indiana
  - St. Joseph Hospital, Lexington, Kentucky
  - Union Memorial Hospital, Baltimore, Maryland
  - St. Mary's Duluth Clinic Regional Heart Center, Duluth, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Our Lady of Lourdes Medical Center, Cherry Hill, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - Wake Medical Center, Raleigh, North Carolina
  - The Carl & Edyth Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Presbyterian University of Pennsylvania Medical Center, Philidelphia, Pennsylvania
  - Fletcher Allen Health Care, Burlington, Vermont
  - St. Mary's Medical Center, Huntington, West Virginia
- Belgium (4):
  - Imelda Ziekenhuis, Bonheiden
  - Universitair Ziekenhuis Gent, Ghent
  - Virga Jesse Ziekenhuis, Hasselt
  - H-Hartziekenhuis Roeselare-Menen vzw, Roeselare
- France (3):
  - Centre Hôpital Universitaire Rangueil, Toulouse, Cedex 9
  - Hospitaux du Haut Leveque, Pessac, Cedex
  - Clinique Pasteur, Toulouse
- Germany (3):
  - Kerckhoff Heart and Thoraxcenter, Bad, Nauheim
  - Herz-Kreislauf-Zentrum Segeberger Kliniken GmbH, Bad Segeberg
  - Universitaetsklinikum Heidelberg, Heidelberg
- P. Stradins University Hospital, Riga, Latvia
- Netherlands (3):
  - Catharina Ziekenhuis, Eindhoven
  - Acadmisch Ziekehus, Maastricht
  - Haga Ziekenhuis locatie Leyweg, The Hague
- Hospital Clinico Y Provincial, Barcelona, Spain

REFERENCES:
- [Derived] Wang JC, Carrie D, Masotti M, Erglis A, Mego D, Watkins MW, Underwood P, Allocco DJ, Hamm CW. Primary endpoint results of the OMEGA Study: One-year clinical outcomes after implantation of a novel platinum chromium bare metal stent. Cardiovasc Revasc Med. 2015 Mar;16(2):65-9. doi: 10.1016/j.carrev.2014.12.007. Epub 2014 Dec 23. PMID 25576273

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OMEGA™ Monorail Coronary Stent System
Started | 328
Completed | 328
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | OMEGA™ Monorail Coronary Stent System
Number analyzed (Participants) | 328
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.46 (11.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106
  Male | 222
Race/Ethnicity, Customized [Number; unit: participants]
  Black, of African heritage | 9
  Caucasian | 254
  Hispanic or Latino | 2
  Other | 2
  Not disclosed | 61
Region of Enrollment [Number; unit: participants]
  France | 55
  United States | 104
  Spain | 39
  Belgium | 37
  Netherlands | 39
  Latvia | 23
  Germany | 31
Cardiac History [Number; unit: participants] — Note: A single participant could potentially experience multiple categories listed below.
  participants
    Previous Myocardial Infarction | 96
    History of CABG | 15
    History of PCI | 95
    History of CHF | 21
    Stable Angina | 182
    Unstable Angina | 111
    Silent Ischemia | 54
Cardiac Risk Factors [Number; unit: participants] — Note: A single participant could potentially experience multiple categories listed below.
  participants
    Smoking, Ever | 211
    Medically Treated Diabetes | 57
    Hyperlipidemia Requiring Medication | 230
    Hypertension Requiring Medication | 243
    Family History of CAD | 131
Lesion Characteristics: Target Lesion Vessel [Number; unit: participants] — Note: A single participant could potentially experience multiple categories listed below.
  participants
    Left Anterior Descending Artery | 112
    Circumflex Artery | 79
    Right Coronary Artery | 137
Lesion Characteristic: Lesion Location [Number; unit: Lesions] — Note: A single participant could potentially experience multiple categories listed below.
  Lesions
    Proximal | 122
    Mid | 155
    Distal | 37
    Ostial | 14
Lesion Characteristic: Lesion Length [Number; unit: Lesions] — Note: A single participant could potentially experience multiple categories listed below.
  Lesions
    Less than 10 mm | 123
    10 to 20 mm | 172
    Greater than 20 mm | 32
Lesion Characteristics [Number; unit: Lesions] — Note: A single participant could potentially experience multiple categories listed below.
  Lesions
    Tortuosity, Any | 32
    Thrombus | 4
    Calcification, Any | 111
    Ulcer | 21
    Aneurysm | 7
Lesion Characteristic: Pre-Procedure Thrombolysis in Myocardial Infarction (TIMI) Flow [Number; unit: Lesions] — Note: A single participant could potentially experience multiple categories listed below.
  Lesions
    0 (no perfusion) | 0
    1 (penetration with minimal perfusion) | 2
    2 (partial perfusion) | 6
    3 (complete perfusion) | 319
Lesion Characteristics by Quantitative Cornary Angiography [Mean (Standard Deviation); unit: Millimeters]
  Reference Vessel Diameter | 2.77 (0.53)
  Minimum Lumen Diameter | 0.9 (0.38)
  Lesion Length | 12.49 (5.15)
Lesion Characteristic: Percent Diameter Stenosis by QCA [Mean (Standard Deviation); unit: Percent] | 67.41 (11.34)

OUTCOME MEASURES:

1. Primary Outcome: 9-month Target Lesion Failure (TLF) Rate
Description: The primary endpoint is 9-month target lesion failure (TLF) rate, defined as any ischemia-driven revascularization of the target lesion (TLR), Myocardial Infarction (MI) (Q-wave and non-Q-wave) related to the target vessel, or cardiac death.
Time Frame: Nine Month
Population: N=323 (5 patients were not evaluable for the endpoint: Follow-up < 240 days and event-free)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMEGA™ Monorail Coronary Stent System
Number analyzed (Participants) | 323
percentage of participants | 11.5 [8.2 to 15.4]

2. Secondary Outcome: 12 Month Target Lesion Revascularization (TLR) Rate
Description: Any ischemia-driven repeat percutaneous coronary intervention (PCI), to improve blood flow, of the successfully treated target lesion or bypass surgery of the target vessel with a graft distally to the successfully treated target lesion.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day, through 12 months
Population: 12-Month rates: the percentage of patients who experience an event through 365 days post-procedure out of the patients who have either had an event within 365 days post-procedure or who were event-free with last follow-up at least 335 days post-procedure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMEGA™ Monorail Coronary Stent System
Number analyzed (Participants) | 322
percentage of participants | 8.4 [5.6 to 12.0]

3. Secondary Outcome: 12 Month Target Vessel Revascularization (TVR) Rate
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day, through 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMEGA™ Monorail Coronary Stent System
Number analyzed (Participants) | 322
percentage of participants | 9.9 [6.9 to 13.7]

4. Secondary Outcome: 12 Month Target Vessel Failure (TVF) Rate
Description: Target vessel failure is any ischemia-driven revascularization of the target vessel, MI (Q-wave and non-Q-wave) related to the target vessel or death related to the target vessel. For the purposes of this protocol, if it cannot be determined with certainty whether the MI or death was related to the target vessel, it will be considered a TVF.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day, through 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMEGA™ Monorail Coronary Stent System
Number analyzed (Participants) | 322
percentage of participants | 13.8 [10.2 to 18.0]

5. Secondary Outcome: 12 Month Myocardial Infarction (MI)(Q-wave and Non-Q-wave) Rate
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day, through 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMEGA™ Monorail Coronary Stent System
Number analyzed (Participants) | 322
percentage of participants | 4.0 [2.2 to 6.8]

6. Secondary Outcome: 12 Month Cardiac Death Rate
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day, through 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMEGA™ Monorail Coronary Stent System
Number analyzed (Participants) | 322
percentage of participants | 1.2 [0.3 to 3.1]

7. Secondary Outcome: 12 Month Non-cardiac Death Rate
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day, through 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMEGA™ Monorail Coronary Stent System
Number analyzed (Participants) | 322
percentage of participants | 0.6 [0.1 to 2.2]

8. Secondary Outcome: 12 Month All Death Rate
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day, through 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMEGA™ Monorail Coronary Stent System
Number analyzed (Participants) | 322
percentage of participants | 1.9 [0.7 to 4.0]

9. Secondary Outcome: 12 Month Cardiac Death or MI Rate
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day, through 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMEGA™ Monorail Coronary Stent System
Number analyzed (Participants) | 322
percentage of participants | 5.3 [3.1 to 8.3]

10. Secondary Outcome: 12 Month All Death or MI Rate
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day, through 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMEGA™ Monorail Coronary Stent System
Number analyzed (Participants) | 322
percentage of participants | 5.9 [3.6 to 9.1]

11. Secondary Outcome: 12 Month All Death/MI/TVR Rate
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day, through 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMEGA™ Monorail Coronary Stent System
Number analyzed (Participants) | 322
percentage of participants | 14.3 [10.7 to 18.6]

12. Secondary Outcome: 12 Month Stent Thrombosis Rate (Definite or Probable by Academic Research Consortium [ARC] Definitions)
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day, through 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OMEGA™ Monorail Coronary Stent System
Number analyzed (Participants) | 314
percentage of participants | 0.6 [0.1 to 2.3]

13. Secondary Outcome: Periprocedural Endpoints: Technical Success Rate
Description: Technical success: successful delivery and deployment of the study stent to the target vessel, without balloon rupture or embolization. Summarized per attempted study stent.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Number (95% Confidence Interval); unit: percentage of patients
Units Other Than Participants: Stents Attempted
Arm/Group | OMEGA™ Monorail Coronary Stent System
Number analyzed (Participants) | 328
Number analyzed (Stents Attempted) | 337
percentage of patients | 98.5 [96.6 to 99.5]

14. Secondary Outcome: Clinical Procedural Success Rate
Description: Clinical Procedural Success: lesion diameter stenosis < 30% in 2 near-orthogonal projections with TIMI 3 flow, as visually assessed by the physician, without the occurrence of in-hospital MI, TVR, or cardiac death. Summarized per patient.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | OMEGA™ Monorail Coronary Stent System
Number analyzed (Participants) | 328
percentage of patients | 95.4 [92.6 to 97.4]

ADVERSE EVENTS:
Time Frame: Serious and non-serious adverse events were collected from the point of subject enrollment through study completion at 12 months.
Arm/Group | OMEGA™ Monorail Coronary Stent System
Serious Adverse Events (participants affected / at risk) | 108/328
Other Adverse Events (participants affected / at risk) | 118/328
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OMEGA™ Monorail Coronary Stent System (N=328)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 4 (4)
Angina pectoris (Cardiac disorders) | 28 (29)
Angina unstable (Cardiac disorders) | 16 (16)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 5 (5)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 3 (3)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiac asthma (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3 (3)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 4 (4)
Coronary artery thrombosis (Cardiac disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Anal polyp (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (2)
Impaired healing (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 10 (10)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Abdominal wall infection (Infections and infestations) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Blood pressure abnormal (Investigations) | 1 (1)
Cardiac enzymes increased (Investigations) | 1 (1)
Cardiac stress test abnormal (Investigations) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1)
B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery disease (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (2)
Hemiplegia (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Mental status changes (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2)
Renal artery stenosis (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 2 (2)
Intermittent claudication (Vascular disorders) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (2)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OMEGA™ Monorail Coronary Stent System (N=328)
Angina pectoris (Cardiac disorders) | 15 (16)
Coronary artery dissection (Cardiac disorders) | 5 (5)
Haemorrhoids (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 6 (6)
Asthenia (General disorders) | 8 (8)
Fatigue (General disorders) | 4 (5)
Non-cardiac chest pain (General disorders) | 13 (13)
Vessel puncture site haemorrhage (General disorders) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (9)
Dizziness (Nervous system disorders) | 5 (6)
Headache (Nervous system disorders) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hypertension (Vascular disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Investigator shall have the right to publish the results, provided that before publishing, Institution and Investigator shall submit copies of any proposed publication or presentation to Sponsor for review at least sixty (60) days in advance of submission for publication or presentation to a publisher or other third party. Sponsor reserves the right to delete any confidential information or other proprietary information of Sponsor from the proposed publication or presentation.